CLINICAL TRIAL: NCT02528721
Title: Clinical Validation Study to Evaluate Presence of H. Pylori With 13C-Urea Breath Test Using the BreathID® Hp Lab System Compared to Biopsy Results
Brief Title: Exalenz Lab Mode System Compared to Biopsy for H.Pylori Detection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DM2-HP-0715
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Diagnosis Subjects (Experimental): Patients with clinical indication for H.pylori infection
  Interventions: Device: Dual Mode BreathID Hp System
- Post Therapy Subjects (Experimental): Patients wishing to confirm eradication of initially diagnosed H.pylori infection that are after treatment within the last 6 months
  Interventions: Device: Dual Mode BreathID Hp System

INTERVENTIONS:
Device: Dual Mode BreathID Hp System — The Dual Mode Breath ID Hp System consists of breath collection bags, a 13C-labelled substrate (urea) and a breath analyzer device
  Other Names: Hp™ TWO; Dual Mode BreathID® Hp

SUMMARY:
The Exalenz Dual Mode BreathID® Hp System comprised of IDkit: Hp™ TWO and the Dual Mode BreathID® Hp test device will be used to perform a urea breath test in the initial diagnosis and post treatment monitoring of H.pylori infection in adult patients and its results will be compared to biopsy results.

DETAILED DESCRIPTION:
Patients undergoing esophagogastroduodenoscopy (EGD) for initial diagnosis of H.pylori infection or post therapy confirmation of eradication will be eligible to participate in the trial. Two sets of biopsies will be taken: one set for histological analysis and one set for rapid urease test (RUT) analysis. The two results will be used as a gold standard composite score in determining the presence of H.pylori bacteria in the stomach. The Urea Breath Test (UBT) using the Exalenz Dual Mode BreathID Hp System will also be performed within a week of the biopsy. The outcome of the UBT will be compared to composite score of the biopsy and the accuracy of the UBT will be evaluated. The UBT will be performed using breath collection bags, where the subject will be asked to breathe into the bags before and after ingestion of the 13C-labelled urea.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have the ability and willingness to sign the Informed Consent Form.
* Present with clinical indication of H. pylori and a candidate for upper endoscopy

For Initial Diagnosis arm:

• Symptomatic patients naïve to H.pylori treatment in the past 18 months

For Post-Therapy arm:

* Documented biopsy with positive outcome prior to eradication therapy (including method of determination)
* Documented eradication therapy within the past 6 months and completed at least 6 weeks prior to UBT

Exclusion Criteria:

* Participation in other interventional trials.

  * Antibiotics and/or Bismuth preparations within four (4) weeks prior to breath test.
  * PPI or H2 blockers within two (2) weeks prior to breath test.
  * Pregnant or breastfeeding women.
  * Allergy to test substrates.
  * Patient did not fast for the hour prior to the UBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Del Sol Research Management, Tucson, Arizona
  - Ventura Clinical Trials, Ventura, California
  - Innovative Clincal Research, Lafayette, Colorado
  - Palmetto Research, Hialeah, Florida
  - Hope Clinical Research, Kissimmee, Florida
  - Metropolitan Gastro Group, Chevy Chase, Maryland
  - Gasrtrenetrology Associates of Western Michigan, West Michigan Clinical Research Center, Wyoming, Michigan
  - Digestive Disease Care, New Hyde Park, New York
  - Great Lakes Medical Research, Willoughby, Ohio
  - Innovative Clinical Research, Rapid City, South Dakota
  - Digestive Disease Center of South Texas, P.L.L.C, San Antonio, Texas
- Israel (2):
  - Barzilai Medical center, Ashkelon
  - Assaf Harofe Medical Center, Tzrifin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Initial Diagnosis Subjects | Post Therapy Subjects
Started | 203 | 79
Completed | 196 | 76
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Diagnosis Subjects | Post Therapy Subjects | Total
Number analyzed (Participants) | 196 | 76 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (14.94) | 49.0 (15.53) | 48.64 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 48 | 164
  Male | 80 | 28 | 108

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity is Described as the Accuracy of the Breath Test in Detecting H.Pylori Infection Compared to Biopsy
Description: Sensitivity of urea breath test with Dual Mode Breath Hp System in accurately detecting presence of H.pylori infection as compared to composite biopsy result
Time Frame: 9 months
Population: According to the FDA Guidelines, if there is a discrepancy between the histology and the rapid urease test results ("composite reference standard"), the subject is considered "unevaluable" and thus not included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percent positive agreement
Arm/Group | Initial Diagnosis Subjects | Post Therapy Subjects
Number analyzed (Participants) | 179 | 68
Percent positive agreement | 98.32 [95.18 to 99.65] | 98.53 [92.08 to 99.96]

2. Primary Outcome: Specificity as Described as the Accuracy of the Breath Test in Detecting Absence of H.Pylori Infection Compared to Biopsy
Description: Specificity of urea breath test with Dual Mode Breath Hp System in accurately detecting lack of presence of H.pylori infection as compared to composite biopsy result
Time Frame: 9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent negative agreement
Arm/Group | Initial Diagnosis Subjects | Post Therapy Subjects
Number analyzed (Participants) | 179 | 68
Percent negative agreement | 97.9 [93.99 to 99.57] | 100 [93.51 to 100]

3. Primary Outcome: Overall Agreement in Determining Presence or Absence of H.Pylori Infection Compared to Biopsy
Description: Overall Agreement of urea breath test with Dual Mode Breath Hp System in accurately detecting presence of H.pylori infection as compared to composite biopsy result
Time Frame: 9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent overall agreement
Arm/Group | Initial Diagnosis Subjects | Post Therapy Subjects
Number analyzed (Participants) | 179 | 68
Percent overall agreement | 98.33 [95.21 to 99.65] | 100 [94.72 to 100]

ADVERSE EVENTS:
Arm/Group | Initial Diagnosis Subjects | Post Therapy Subjects
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/79
Other Adverse Events (participants affected / at risk) | 4/203 | 1/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Diagnosis Subjects (N=203) | Post Therapy Subjects (N=79)
Cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cyst discovered on epiglottis during standard EGD procedure
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastric ulcer discovered during EGD procedure
Nausea (General disorders) | 2 (2) | 0 (0) — Nausea experienced for two minutes after drinking test substrate
Lightheadedness (General disorders) | 0 (0) | 1 (1) — Lightheadedness due to fasting for standard EGD procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less